CLINICAL TRIAL: NCT03511157
Title: Walking Capacity of Patients With Claudication in Lower Extremities Following Ischemic Preconditioning
Brief Title: Ischemic Preconditioning Claudication Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Matthew Durand, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00031772
Record Dates: First submitted 2018-04-09; First posted 2018-04-27 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Intermittent Claudication; Ischemia Vascular; Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: ischemic preconditioning
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — Ischemic Preconditioning; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Preconditioning (Experimental): A standard blood pressure cuff will be placed on the right or left thigh, depending on the affected side, to occlude blood flow. The cuff will be inflated to 225 mmHg to prevent blood flow. Each session will consist of 4 cycles of 5 minute IPC applications, followed by 5 minutes of reperfusion for a total of 35 minutes.
  Interventions: Other: Ischemic Preconditioning
- Control (Sham Comparator): The sham intervention protocol will be identical to the IPC protocol except blood flow to the affected leg is unchanged as cuff pressure will be raised to between the venous and diastolic pressures
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Ischemic Preconditioning — See Ischemic Preconditioning Experimental group description
  Arms: Ischemic Preconditioning
Other: Control Group — See Control group description
  Arms: Control

SUMMARY:
This study proposes ischemic preconditioning (IPC) as a novel intervention to improve walking distance in patients with intermittent claudication.

DETAILED DESCRIPTION:
This study proposes ischemic preconditioning (IPC) as a novel intervention to improve walking distance in patients with intermittent claudication. Peripheral arterial disease (PAD) is a circulatory condition in which large supply blood vessels narrow, reducing oxygen and nutrient distribution to peripheral tissues. IPC protects against tissue damage caused by ischemia and can improve functional capacity in patients recovering from stroke; however, the benefit of ischemic preconditioning in patients with peripheral arterial disease remains unclear.

The investigators predict that ischemic preconditioning (IPC) will delay claudication onset time (COT), increase peak walking time (PWT) and improve muscle strength in patients with intermittent claudication.

The investigators will determine whether IPC improves claudication onset time (COT) and peak walking time (PWT) in patients with intermittent claudication. A motorized treadmill will be employed to assess COT and PWT.

The investigators will determine whether IPC can improve muscle strength and time to pain onset in the affected leg of patients with intermittent claudication. These metrics will be assessed quantitatively using a Biodex™ dynamometer.

ELIGIBILITY:
Inclusion Criteria:

1. between ages of 18-80
2. able to give informed consent
3. presence of vascular disease with intermittent claudication

Exclusion Criteria:

1. age < 18 or >80
2. unable to give informed consent
3. presence of vascular disease with leg pain at rest, ischemic ulceration, or gangrene
4. pregnancy
5. unable to walk on a treadmill
6. unable to perform or tolerate ischemic preconditioning
7. unable to follow commands
8. exercise capacity limited by symptoms of angina, congestive heart failure, chronic obstructive pulmonary disease, or arthritis to be determined by PI
9. patients who have undergone vascular surgery or endovascular surgery in the previous year on the affected leg
10. history of major lower extremity amputation
11. history of major psychiatric disorder
12. history of uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Peak walking time | 2 weeks
  Subjects will be placed on a motorized treadmill and peak walking time will be recorded in seconds.

SECONDARY OUTCOMES:
Muscle Fatigue | 2 weeks
  Subjects will perform muscle contractions for muscle groups of interest (knee extensors/flexors and dorsiflexors/plantarflexors). Contractions will be measured in newton-meters. The duration will be determined by the time subjects first feel pain and when the pain becomes too great to continue. The investigators will provide subjects with visual feedback on the monitor throughout the testing.
Claudication onset time | 2 weeks
  Subjects will be placed on a motorized treadmill and claudication onset time will be recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No